CLINICAL TRIAL: NCT06462196
Title: Natural History of Depression, Bipolar Disorder and Suicide Risk
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001874; 001874-M
Record Dates: First submitted 2024-06-14; First posted 2024-06-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Behavioral Symptoms; Suicide; Self-Injurious Behavior; Sensory System Agents; Analgesics; Peripheral Nervous System Agents; Physiological Effects of Drugs; Anesthetics, Dissociative; Anesthetics, General; Anesthetics; Central Nervous System Depressants; Excitatory Amino Acid Antagonists; Excitatory Amino Acid Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Ketamine; Depression, Unipolar; Depressive Symptoms; Treatment Resistant Depression; Major Depressive Disorder; Depression, Bipolar
Keywords: Neurobiology; Suicide; Major Depressive Disorder; Bipolar Disorder; Biomarkers; Suicide Risk; Treatment Resistant Depression
MeSH Terms: conditions — Behavioral Symptoms; Suicide; Self-Injurious Behavior; Depressive Disorder; Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bipolar Disorder: Individuals with Bipolar Disorder
- Major Depressive Disorder: Individuals with Major Depressive Disorder
- Suicide Risk: Individuals at an elevated suicide risk

SUMMARY:
Mood disorders, such as depression and bipolar disorder, are difficult to treat. One reason is that there are no objective ways to measure how these disorders affect the body and respond to different treatments. In this study, researchers want to perform tests on people undergoing clinical care for mood disorders. The purpose is to understand the experience of receiving treatment for depression, bipolar disorder, and suicide risk. We also hope that this study will help us to predict which medications will improve thoughts of suicide.

People 18 years or older who are receiving treatment for depression, bipolar disorder, or suicide risk may take part in this study. Participants must have also been enrolled in protocol 01-M-0254.

This study will be conducted at the NIH Clinical Center in Bethesda, MD. The study typically lasts up to 12 weeks, but may last longer if a participant s treatment continues past that time.

Participants will have weekly interviews and questionnaires while they are being treated for their mood disorder. Other tests are optional and include psychological testing, blood draws, sleep tests, and imaging scans. These will be done at the start and the end of research participation.

DETAILED DESCRIPTION:
Study Description:

This proposal would collect systematic data on individuals undergoing personalized treatments for depression, bipolar disorder and suicide risk within the Experimental Therapeutics and Pathophysiology Branch (ETPB). The ETPB recruits individuals with treatment-resistant mood disorders from around the country. After research participation, they are often offered a course of standard treatment, tailored to clinical needs, for clinical stabilization and discharge back to non-NIH clinicians. This protocol would allow for clinical ratings in-person and remotely throughout clinical standard treatments, as well as neurobiological procedures at baseline and study termination to identify potential clinical and demographic predictors and biomarkers of treatment response.

Objectives:

The primary objective is to identify predictors of antidepressant treatment response.

The secondary and tertiary objectives are to identify predictors of suicide ideation response to treatment, and biomarkers of antidepressant response to treatment, respectively.

Endpoints:

Primary Endpoint: Score on the Montgomery Asberg Depression Rating Scale

Secondary Endpoint: Score on the Scale for Suicidal Ideation

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Signed consent for Protocol 01-M-0254: The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers
* Age 18 years or older
* Able to provide informed consent
* Able to read and write English

EXCLUSION CRITERIA:

* Unstable medical conditions in the opinion of the investigator that would preclude participation in outpatient or inpatient treatment.
* Pregnancy
* Participation in the Protocol 01-M-0254: The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers, as a healthy volunteer.
* Participants with a history of DSM-IV substance or alcohol abuse or dependence, or DSM-5 substance use disorder (except for caffeine, nicotine, or cannabis), or moderate to severe alcohol use disorder, within the preceding three months. In addition, participants who are currently using drugs (except for caffeine, nicotine, or cannabis) must not have used illicit substances or known drugs of abuse in the two weeks prior to consent and must have a negative drug urine test (except for prescribed benzodiazepines or stimulants) prior to enrolling in the study. Cannabis use is exclusionary if the use is daily, or if participants are unable to abstain during the study, or if function of daily life is impaired by use as determined by a clinician.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with depression, bipolar disorder, and individuals at elevated suicide risk.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Score on Montgomery Asberg Depression Rating Scale | Weekly
  Depression rating scale

SECONDARY OUTCOMES:
Score on Scale for Suicide Ideation | Weekly
  Scale for rating suicide ideation

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D Ballard, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and research ratings, multi-modal MRI images, MEG scans, sleep studies, physiological, behavioral, and phenotypic data collected during the study, after deidentification.
Supporting Information: SAP
Time Frame: Starting within 1 year of completion of the study
Access Criteria: Participants data will only be shared if they have opted into the data share agreement. Data deposited into repositories will not be subject to any access, distribution, or reuse limitation beyond the standard procedures of the repository. Data will be uploaded to repositories listed in our NIH Intramural Research Program (IRP) Data Management and Sharing Plan. There are no restrictions on subsequent access, distribution, or reuse once the data is placed in a repository. The Branch Chief will review requests and access will need to be approved by the NIMH/DIRP SD and OCD NIMH and the NIH IRB.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001874-M.html